CLINICAL TRIAL: NCT06377410
Title: A Randomised, Open Label, Interventional Study Evaluating the Efficacy & Safety of Dry Powder Ivy Extract (Syrup Prospan) Versus NAC Among COPD Patients (SyProNAC Trial)
Brief Title: Efficacy & Safety of Dry Powder Ivy Extract (Syrup Prospan) Versus NAC Among COPD Patients
Acronym: SyProNAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FF-2023-433
Record Dates: First submitted 2024-03-31; First posted 2024-04-22 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participant with stable COPD who received Syrup prospan (Active Comparator): Participant who fulfiled inclusion criteria with stable COPD and received Syrup prospan for 1 month
  Interventions: Drug: Syrup Prospan
- Participant with stable COPD who received N-Acetylcysteine (Active Comparator): Participant who fulfiled inclusion criteria with stable COPD and received SN-Acetylcysteine for 1 month
  Interventions: Drug: N-Acetylcysteine

INTERVENTIONS:
Drug: Syrup Prospan — Participant with stable COPD who received Syrup prospan for 1 month
  Arms: Participant with stable COPD who received Syrup prospan
Drug: N-Acetylcysteine — Participant with stable COPD who received N-Acetylcysteine for 1 month
  Arms: Participant with stable COPD who received N-Acetylcysteine

SUMMARY:
As the third global leading cause of death, Chronic Obstructive Pulmonary Disease (COPD) affects more than 300 million people worldwide. These patients suffer from 0.5-3.5 exacerbations per year on average. Each exacerbations dampened their health status as well as quality of life, not to mention a great burden to our healthcare system. Those partially treated or prolonged exacerbations would subsequently lead to unfavorable disease progression. Hence a holistic approach in managing each exacerbations is very crucial.

Mucus hypersecretion in COPD patients plays a pivotal role in acute exacerbations and associated with unfavorable outcomes. These exacerbations comes with sputum increment as much as its purulence. Mucolytics are believed to to ease patient to expectorate and benefits them from tip into an exacerbations or even the consequent hospitalisation.

Mucolytics work by reducing sputum viscosity hence improved its expectoration. N-acetylcysteine (NAC) is a mucolytic with antioxidant and anti-inflammatory properties, commonly used in practice among COPD patients. Meanwhile, Syrup Prospan is ivy leaf preparations, obtained as extracts from leaves of the plant Hedera helix L. It is widely used over-the-counter cough remedy containing saponins which are believed to have expectorant properties. Studies show evidence of antispasmodic, bonchodilating, anti-inflammatory and antitussive properties and its usage is authorised by the European Medicines Agency .

DETAILED DESCRIPTION:
Hypothesis

1. Syrup Prospan is non inferior to NAC - no significant difference of cough symptoms and its impact on daily activities, health related quality of life, as well as lung function test at 30 days of treatment
2. Patients received Syrup Prospan has higher satisfaction score compared to N-Acetylcysteine

This is a randomised, open label, interventional study evaluating the efficacy and safety of dry powder Ivy Extract (Syrup Prospan) versus NAC among COPD patients. Randomization 1:1 to received either N.Acetylcysteine 600 mg BD or Syrup Prospan 7.5mls BD (Block randomization)

The study will be conducted from April 2024 to November 2026 This is a prospective interventional study conducted on COPD patients under the Respiratory Unit, Department of Internal Medicine in HCTM, who qualified both the inclusion and exclusion criteria. Patients will be briefed about this study.

Subsequently, consent will be obtained from those who are agree to participate from the patient him/herself.

Participants' will be assessed first with several modalities particularly spirometry, CAT score, McGill COPD Quality of Life and Cough and Sputum Assessment Questionnaire (CASA-Q) prior to the commencement of treatment.Participants will be seen on Day 15 to evaluate patients' adherence, compliance as well as adverse effect. Then patients will be assessed again on Day 30 of treatment with the same set of evaluation tools as in the beginning of the study.

In order to calculate the required sample size, we will employ the Cohen's d formula for estimating the effect size (Cohen, 1988) [19]. The formula is given as

Where d is the Cohen's effect size, M1 and M2 are the mean for the first and second group, and SD1 and SD2 are the standard deviation for the first and second group respectively.

Based on a previous study which employs the CAT score to assess the efficacy of NAC in patients with COPD, the mean and standard deviation for before and after treatment are given as:

Before treatment: 23.46 ± 3.66 After treatment: 20.38 ± 5.78

Hence, this give the values of M1 = 23.46 and M2 = 20.38, and SD1 =3.66 and SD2 = 5.78 that can use to estimate the effect size using the formula above.

Therefore, it gives an estimated effect size of 0.637 which is considered to be a medium effect size.

With a power of 80% and a level of significance of 5% for detecting an effect size of 0.637, we calculate the required sample size using an online sample size calculator for comparing paired differences. It gives at a value of 23 participants for each group which mean the required number of participants is 46.

Additional of 20% samples is recruited to avoid missing data due to withdrawal or drop out. Therefore, a total of minimum 55 patients will be recruited for this study. However, we aim to recruit 100 patients for our study where the treatment is given to equal number of participants in each group.

ELIGIBILITY:
Inclusion Criteria:

* Participants with documented post bronchodilator FEV1/FVC < 70 or <LLN
* Age 40 years and above
* Able to perform spirometry
* Participant with Stable COPD based on GOLD 2023 strategy

Exclusion Criteria:

* Diagnosis of other chronic lung diseases: Asthma, Asthma-COPD Overlap, Interstitial Lung Disease, Bronchiectasis, Lung Cancer
* Participants with contraindication for spirometry: recent cardiac complications, major surgery, severe advanced respiratory disease, or those with cognitively or neurologically impairment
* Hypersensitivity to acetylcysteine or any component of the formulation
* Hypersensitivity to dry powder ivy extract
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG (human Chorionic Gonadotropin) laboratory test
* Participant on pre-existing regular mucolytics (at least 1 month prior)
* Illiterate participants

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
To assess cough symptoms and its impact on daily activities using Cough and Sputum Assessment Questionnaire (CASA-Q); scores for each domain range from 0 to 100, with higher scores indicating fewer/less severe symptoms and less impact. | From the time of randomization to the time of the end of study up to 30 days post randomization
  Participants with COPD who received either Syrup Prospan or N-Acetylcysteine

SECONDARY OUTCOMES:
to determine change of Quality of Life using McGill COPD Quality of Life Questionnaire, scores ranged from 0 to 100, with higher scores indicating a better quality of life. | From the time of randomization to the time of the end of study up to 30 days post randomization
  Participants with COPD who received either Syrup Prospan or N-Acetylcysteine
to determine change of Forced Expiratory Volume at 1second (FEV1); in litres/minute using spirometry | From the time of randomization to the time of the end of study up to 30 days post randomization
  Participants with COPD who received either Syrup Prospan or N-Acetylcysteine
to determine change of Forced Vital Capacity in litres/minute using spirometry | From the time of randomization to the time of the end of study up to 30 days post randomization
  Participants with COPD who received either Syrup Prospan or N-Acetylcysteine
to determine adverse effects of Syrup Prospan (in %) | From the time of randomization to the time of the end of study up to 30 days post randomization
  Participants with COPD who received Syrup Prospan
to determine adverse effects of N-Acetylcysteine (in %) | From the time of randomization to the time of the end of study up to 30 days post randomization
  Participants with COPD who received N-Acetylcysteine
To assess satisfaction of treatment using the 5 point Likert Scale (1- Not Satisfied, 5 - Most Satisfied) | From the time of randomization to the time of the end of study up to 30 days post randomization
  Participants with COPD who received either Syrup Prospan or N-Acetylcysteine

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Faisal Abdul Hamid, MBBS (IIUM), Principal Investigator — National University of Malaysia
Locations (2):
- Malaysia (2):
  - National University of Malaysia, Faculty of Medicine, Cheras, Kuala Lumpur
  - National University of Malaysia, Cheras, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] GBD 2017 DALYs and HALE Collaborators. Global, regional, and national disability-adjusted life-years (DALYs) for 359 diseases and injuries and healthy life expectancy (HALE) for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1859-1922. doi: 10.1016/S0140-6736(18)32335-3. PMID 30415748
- [Result] Seemungal TA, Hurst JR, Wedzicha JA. Exacerbation rate, health status and mortality in COPD--a review of potential interventions. Int J Chron Obstruct Pulmon Dis. 2009;4:203-23. doi: 10.2147/copd.s3385. Epub 2009 Jun 11. PMID 19554195
- [Result] Donaldson GC, Wedzicha JA. COPD exacerbations .1: Epidemiology. Thorax. 2006 Feb;61(2):164-8. doi: 10.1136/thx.2005.041806. PMID 16443707
- [Result] Donaldson GC, Law M, Kowlessar B, Singh R, Brill SE, Allinson JP, Wedzicha JA. Impact of Prolonged Exacerbation Recovery in Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2015 Oct 15;192(8):943-50. doi: 10.1164/rccm.201412-2269OC. PMID 26151174
- [Result] Garrard J, Rolnick SJ, Nitz NM, Luepke L, Jackson J, Fischer LR, Leibson C, Bland PC, Heinrich R, Waller LA. Clinical detection of depression among community-based elderly people with self-reported symptoms of depression. J Gerontol A Biol Sci Med Sci. 1998 Mar;53(2):M92-101. doi: 10.1093/gerona/53a.2.m92. PMID 9520914
- [Result] Poole P, Sathananthan K, Fortescue R. Mucolytic agents versus placebo for chronic bronchitis or chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2019 May 20;5(5):CD001287. doi: 10.1002/14651858.CD001287.pub6. PMID 31107966
- [Result] Du Y, Wolf IK, Zhuang W, Bodemann S, Knoss W, Knopf H. Use of herbal medicinal products among children and adolescents in Germany. BMC Complement Altern Med. 2014 Jul 2;14:218. doi: 10.1186/1472-6882-14-218. PMID 24988878
- [Result] Balsamo R, Lanata L, Egan CG. Mucoactive drugs. Eur Respir Rev. 2010 Jun;19(116):127-33. doi: 10.1183/09059180.00003510. PMID 20956181

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT06377410/Prot_SAP_ICF_000.pdf